CLINICAL TRIAL: NCT06867107
Title: An Open-Label Long-Term Follow-up Study of SAT-3247 in Patients With Duchenne Muscular Dystrophy (DMD) That Participated in SAT-3247-CL-101
Brief Title: A Long-term Follow-up Study for Participants That Completed the SAT-3247-CL-101 Study
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Satellos Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAT-3247-LT-001
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: muscle regeneration; SAT-3247
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: open-label study of 60 mg SAT-3247 in 5-days on/2-days off (i.e., weekday dosing) regimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): SAT-3247 60 mg administered orally in a 5-days on/2-days off (weekday) dosing regimen
  Interventions: Drug: SAT-3247

INTERVENTIONS:
Drug: SAT-3247 — AAK1 inhibitor

SUMMARY:
This is an open-label long-term safety and efficacy study of orally administered SAT-3247 in patients with DMD that previously participated in SAT-3247-CL-101.

The study will assess the long-term safety, tolerability and potential efficacy of long-term dosing of 60 mg of orally administered SAT-3247 in a 5-days on/2-days off (i.e. weekday dosing) regimen in an open-label design through 11 months- for a total of 12 months of treatment including the duration of the SAT-3247-CL-101 study. The study will enroll up to 10 participants that previously participated in the SAT-3247-CL-101 study.

ELIGIBILITY:
Inclusion Criteria:

* Previously participated in the SAT-3247-CL-101 parent clinical trials.
* Continued status of stable glucocorticosteroid dose or no glucocorticosteroid dose from parent clinical trial.
* Continued stable doses of prescription medicines (excluding glucocorticosteroids) and over-the-counter medicines and/or herbal supplements for supportive care from parent clinical trial.
* Ability to understand the nature of the trial and any hazards of participating.
* Ability to communicate satisfactorily with the investigator and physiotherapist and to participate in and comply with the requirements of the entire trial including scheduled visits, procedures, laboratory tests, questionnaires, wearable devices, and study restrictions.
* Willingness to give written consent or assent (if not of cognitive capacity of consent in the jurisdiction where the study is being conducted) and parent/legal guardian willing to give written consent to participate (if participant is not of cognitive capacity to consent) after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or their delegate.
* All participants, if sexually active, agree to follow the contraception requirements and sperm donation limitations of the trial as described in the protocol.

Exclusion Criteria:

* Presence of acute medical condition, chronic illness or history of chronic illness (other than DMD) sufficient to invalidate the participant's participation in the trial or make it unnecessarily hazardous in the judgment of the investigator.
* Participants expected to require spine surgeries or hospitalizations for non-acute health needs within 12 months.
* Participants with acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea, heartburn) or acute infection (such as influenza) or a significant infection or known inflammatory process at Screening.
* Severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the investigator.
* Development of symptomatic cardiomyopathy since completion of the parent trial.
* Inability to swallow tablets.

  a. Tablets can be split or crushed and stirred into flavored beverages or food (e.g., apple sauce, yogurt) followed by immediate administration.
* Receipt of an investigational product (including prescription medicines and investigational devices) as part of another clinical trial since completion of the parent trial or in the follow-up period of another clinical trial at the time of Screening for this study.

  a. Use of deflazacort or vamorolone in jurisdictions where these are considered investigational as they have not received health authority marketing authorization will not be exclusionary.
* Possibility that the participant will not cooperate with the requirements of the protocol or is unable or unwilling to comply with the study requirements according to investigator's decision.
* Employee, contractors, or consultants of the Sponsor, the CRO, and/or study site or their relatives.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | 11 months
  Incidence, temporal profile, and severity of treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
SAT-3247 effect on fat fraction in biceps brachii | 12 months
  Changes from baseline in intramuscular fat fraction in muscle quantitative magnetic resonance (qMR) in biceps brachii following treatment with SAT-3247.
SAT-3247 effects on muscle force | 12 months
  Changes from baseline in muscle force measurements as determined by dynamometry following treatment.
Potential for improvement in muscle function with treatment of SAT-3247 | 12 months
  Changes from baseline in Performance of Upper Limb (PUL2.0) assessment following SAT-3247 treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No